CLINICAL TRIAL: NCT00432029
Title: Correlation of Flicker Induced and Flow Mediated Vasodilatation in Patients With Endothelial Dysfunction and Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Wolzt, Medical University of Vienna Department of Clinical Pharmacology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-180506
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus, Type 1; Hypertension; Hypercholesterolemia; Regional Blood Flow
Keywords: Flicker induced vasodilatation; Flow mediated vasodilatation; Forearm blood flow; Retinal vessel diameter; Endothelial dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypertension; Hypercholesterolemia

ARMS (3):
- 1 (Other): IDDM
  Interventions: Procedure: Forearm blood flow measurement, Flow mediated dilation (FMD); Device: Zeiss Retinal Vessel Analyzer (RVA), Stimulation with Flicker-light
- 2 (Other): Hypercholesterolemia and/or Hypertension
  Interventions: Procedure: Forearm blood flow measurement, Flow mediated dilation (FMD); Device: Zeiss Retinal Vessel Analyzer (RVA), Stimulation with Flicker-light
- 3 (Other): age/sex matched healthy control subjects
  Interventions: Procedure: Forearm blood flow measurement, Flow mediated dilation (FMD); Device: Zeiss Retinal Vessel Analyzer (RVA), Stimulation with Flicker-light

INTERVENTIONS:
Procedure: Forearm blood flow measurement, Flow mediated dilation (FMD) — Forearm blood flow measurement: baseline 1 min, 3 min after inflation of cuff, 4 min after 0.8mg Nitroglycerin
Device: Zeiss Retinal Vessel Analyzer (RVA), Stimulation with Flicker-light — Stimulation with Flicker-light: 1 min, measurement without flickering light 4 min after 0.8 mg Nitroglycerin

SUMMARY:
A couple of studies have shown that illuminating the eye with diffuse flickering light is accompanied by an increase of retinal vessel diameters, optic nerve head blood flow and retinal blood flow. We have recently used this visual stimulation technique as a new and powerful tool for the non-invasive investigation of vascular reactivity. Additionally, we could show that this response is diminished in patients with vascular pathologies and that the response is dependent on nitric oxide, indicating that flicker induced vasodilatation may reflect endothelial dysfunction and may be a new approach to test endothelial function in vivo.

One of the most widely used method for the assessment of endothelial function is flow mediated dilatation (FMD). FMD has been shown to give a reliable estimate of vascular function in vivo. In the present study, we set out to compare the standard method for the evaluation of endothelial function, FMD, to flicker induced vasodilatation in the retina.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetic retinopathy:

* Men and women aged > 18 years.
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant.
* Inclusion criteria of patients are insulin dependent diabetes mellitus (IDDM) with non or mild non-proliferative diabetic retinopathy. Patients with no signs of diabetic retinopathy (level 1) or patients with one or more microaneurysms (level 2) will be included. Level of diabetic retinopathy will be assessed according to the criteria defined in the AREDS-study.(1991)
* serum cholesterol < 250 mg/dl (treated or untreated)

Patients with mild hypertension and/or hypercholesterinemia:

* Men and women aged > 18 years.
* mild essential hypertension defined as a blood pressure meeting the criterion of hypertension grade 1 of the World Health Organisation blood pressure classification
* systolic blood pressure between 140 and 159 mmHg and diastolic blood pressure between 90 and 99 mmHg and/or
* serum cholesterol > 250 mg/dl
* blood pressure will be measured at two different occasion in a sitting positions

Healthy subjects:

* Men and women aged > 18 years.
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* normal ocular findings
* serum cholesterol < 200 mg/dl
* systolic blood pressure between 110mmHg and 140mmHg
* diastolic blood pressure < 90 mmHg

Exclusion Criteria:

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* other ocular pathologies than diabetic retinopathy level 1 or 2
* History or family history of epilepsy
* Ametropy greater or equal than 3 dpt
* systolic blood pressure < 100mmHg
* diastolic blood pressure < 75mmHg
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Retinal vessel diameters (Retinal vessel analyzer) | 8 min
Forearm Blood Flow | 8 min

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pemp B, Garhofer G, Weigert G, Karl K, Resch H, Wolzt M, Schmetterer L. Reduced retinal vessel response to flicker stimulation but not to exogenous nitric oxide in type 1 diabetes. Invest Ophthalmol Vis Sci. 2009 Sep;50(9):4029-32. doi: 10.1167/iovs.08-3260. Epub 2009 Apr 15. PMID 19369238